CLINICAL TRIAL: NCT00005584
Title: Prospective Controlled Trial in Clinical Stages I-II Supradiaphragmatic Hodgkin's Disease: Evaluation of Treatment Efficacy, (Long Term) Toxicity and Quality of Life in Two Different Prognostic Subgroups
Brief Title: Combination Chemotherapy With or Without Radiation Therapy in Treating Patients With Hodgkin's Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Lymphoma Study Association (Other); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-20982; FRE-FNCLCC-98014 (Other: FRE-FNCLCC); GELA-H9 (Other: GELA)
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; adult lymphocyte predominant Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; ABVD protocol; Epirubicin; Prednisone; Vinblastine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: ABVD regimen
Drug: BEACOPP regimen
Drug: epirubicin hydrochloride
Drug: prednisone
Drug: vinblastine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy with radiation therapy may kill more cancer cells. It is not yet known which combination chemotherapy regimen is most effective in treating Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of different regimens of combination chemotherapy with or without radiation therapy in treating patients who have Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the late toxicity of 6 courses of epirubicin, bleomycin, vinblastine, and prednisone (EBVP) followed by involved-field radiotherapy (IF-RT) (36 Gy) vs IF-RT (20 Gy), vs no IF-RT (closed to accrual as of 6/2002) in patients with supradiaphragmatic Hodgkin's lymphoma, favorable prognosis, and complete remission (CR) or CR unconfirmed after completion of chemotherapy. (Favorable prognosis group [group 1] closed to accrual as of 4/28/04.)
* Compare 6 courses of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) vs 4 courses of ABVD vs 4 courses of cyclophosphamide, doxorubicin, vincristine, bleomycin, etoposide, procarbazine, and prednisone (BEACOPP) followed by IF-RT, with respect to overall survival and late treatment-related toxicity, in patients with supradiaphragmatic Hodgkin's lymphoma and unfavorable prognosis. (Unfavorable prognosis group [group 2] closed to accrual as of 9/2002.) (Favorable prognosis group [group 1] closed to accrual as of 4/28/04.)
* Maintain the failure-free survival and relapse-free survival rates that were reached in the previous EORTC studies (H5 to H8), with a reduction in acute and delayed side effects of the treatment, in particular that of severe late radiotherapy and chemotherapy-related toxicity.
* Compare the quality of life, overall survival, treatment quality control, and duration of treatment in patients with favorable (closed to accrual as of 4/28/04) or unfavorable (closed to accrual as of 9/2002) prognoses treated with these regimens.
* Determine the efficacy of conservative therapy comprised of observation until disease progression (DP) and administration of IF-RT at the time of DP in patients with lymphocyte-predominant Hodgkin's lymphoma, nodular subtype (nodular paragranuloma).

OUTLINE: This is a randomized, multicenter study.

Patients with classical Hodgkin's lymphoma are assigned to 1 of 2 randomized groups. (Group 2 [unfavorable prognosis] closed to accrual as of 9/2002.) (Group 1 [favorable prognosis] closed to accrual as of 4/28/04.) Patients with lymphocyte-predominant Hodgkin's lymphoma are assigned to the nonrandomized group.

Randomized groups

* Patients are stratified by prognosis (favorable vs unfavorable). Patients are assigned to 1 of 2 treatment groups based on prognosis. (Group 2 [unfavorable prognosis] closed to accrual as of 9/2002.) (Group 1 [favorable prognosis] closed to accrual as of 4/28/04.)

  * Group 1 (favorable prognosis) (closed to accrual as of 4/28/04): Patients receive epirubicin IV over 5 minutes, bleomycin intramuscularly (IM) (or IV if necessary), and vinblastine IV on day 1 and oral prednisone on days 1-5. Treatment repeats every 3 weeks for 6 courses. Patients are then assigned to 1 of 3 involved-field radiotherapy (IF-RT) groups based on response to chemotherapy:

    * Group A (complete remission (CR) or CR unconfirmed [CRu]) Patients are randomized to 1 of 3 radiotherapy arms. (Arm III closed to accrual as of 6/2002.)

      * Arm I (36 Gy): Patients undergo IF-RT 5 days a week for 3.5 weeks.
      * Arm II (20 Gy): Patients undergo IF-RT 5 days a week for 2 weeks.
      * Arm III (closed to accrual as of 6/2002): Patients undergo no IF-RT.
    * Group B (partial remission [PR]): Patients undergo IF-RT 5 days a week for 3.5 weeks and boost radiotherapy.
    * Group C (stable disease or disease progression [DP]): Patients receive no IF-RT and are taken off study.
  * Group 2 (unfavorable prognosis) (closed to accrual as of 9/2002): Patients are randomized to 1 of 3 treatment arms.

    * Arm I: Patients receive doxorubicin IV over 5 minutes, bleomycin IM (or IV if necessary), vinblastine IV, and dacarbazine IV over 5-10 minutes on days 1 and 15. Treatment repeats every 4 weeks for 6 courses.
    * Arm II: Patients receive chemotherapy as in arm I. Treatment repeats every 4 weeks for 4 courses.
    * Arm III: Patients receive cyclophosphamide IV and doxorubicin IV over 5 minutes on day 1, vincristine IV and bleomycin IM (or IV if necessary) on day 8, etoposide IV over a minimum of 30 minutes on days 1-3, oral procarbazine on days 1-7, and oral prednisone on days 1-14. Treatment repeats every 3 weeks for 4 courses.

Patients on all arms who achieve CR or CRu undergo IF-RT 5 days a week for 3 weeks. Patients who achieve PR undergo IF-RT 5 days a week for 3.5 weeks and boost radiotherapy.

* Groups 1 and 2 (group 2 closed to accrual as of 9/2002) (group 1 closed to accrual as of 4/28/04): IF-RT begins within 3-4 weeks after completion of the last course of chemotherapy.

Nonrandomized group

* Patients with completely resected stage I disease undergo observation until DP and undergo IF-RT after documentation of DP. Patients with stage II or incompletely resected stage I disease undergo IF-RT immediately.

Quality of life is assessed before starting study therapy, immediately after completion of study, and then annually for 10 years.

Patients are followed at 2, 4, 6, 9, and 12 months; every 4 months for 1 year; every 6 months for 3 years; and then annually thereafter.

PROJECTED ACCRUAL: A total of 903 patients (group 1) will be accrued for this study within 7.7 years. A total of 723 patients (group 2) will be accrued for this study within 3.8 years. (Group 2 [unfavorable prognosis] closed to accrual as of 9/2002.) (Group 1 [favorable prognosis] closed to accrual as of 4/28/04.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Randomized groups: Histologically proven previously untreated stage I or II supradiaphragmatic Hodgkin's lymphoma

  * No prior staging laparotomy
  * Favorable (closed to accrual as of 4/28/04) or unfavorable (closed to accrual as of 9/2002) prognosis
* Nonrandomized group: Histologically proven lymphocyte-predominant Hodgkin's lymphoma, nodular subtype (nodular paragranuloma)

  * Stage I with complete or incomplete resection OR
  * Stage II

PATIENT CHARACTERISTICS:

Age:

* 15 to 70

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No severe cardiac disease that would interfere with normal life expectancy or study treatment

Pulmonary:

* No severe pulmonary disease that would interfere with normal life expectancy or study treatment

Other:

* No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No severe neurologic or metabolic disease that would interfere with normal life expectancy or study treatment
* No psychologic, familial, socioeconomic, or geographic circumstances that would preclude proper staging or compliance
* HIV negative
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for this malignancy

Chemotherapy

* No prior chemotherapy for this malignancy

Endocrine therapy

* No prior endocrine therapy for this malignancy

Radiotherapy

* No prior radiotherapy for this malignancy

Surgery

* No prior surgery for this malignancy

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1649 (Actual)
Dates: Start 1998-10 (Actual); Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Relapse-free rate | 5 years
  with events defined as lack of CR/CRu at the end of treatment or relapse

SECONDARY OUTCOMES:
Overall Survival | Till withdrawal criteria met
Failure Free Survival | Till withdrawal criteria met
Relapse Free Survival | Till withdrawal criteria met

CONTACTS AND LOCATIONS:
Overall Officials: Jose Thomas, MD, Study Chair — University Hospital, Gasthuisberg; H. Eghbali, MD, Study Chair — Institut Bergonié; E.M. Noordijk, MD, Study Chair — Leiden University Medical Center; Christophe Ferme, Study Chair — Centre Medical de Bligny; Christian Gisselbrecht, MD, Study Chair — Hopital Saint-Louis; Thierry O. Philip, MD, Study Chair — Centre Leon Berard
Locations (121):
- Belgium (10):
  - Sint Augustinus Ziekenhuis, Antwerp
  - A.Z. St. Jan, Bruges
  - C.H.U. Saint-Pierre, Brussels
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
  - Clinique Saint-Pierre, Ottignies
- France (77):
  - Centre Hospitalier Annemasse Bonneville, Ambilly
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Hospital General Robert Ballanger, Aulnay-sous-Bois
  - Hopital Duffaut, Avignon
  - Centre Hospitalier de la Cote Basque, Bayonne
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital de Beziers, Béziers
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - CMC Bligny, Briis-sous-Forges
  - CHU de Caen, Caen
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Regional de Chambery, Chambéry
  - Hopital Fontenoy, Chartres
  - Centre d'Oncologie et de Radiotherapie de Chaumont le Bois, Chaumont
  - Hopital d'Instruction des Armees Percy, Clamart
  - Hopital Antoine Beclere, Clamart
  - Hopital Beaujon, Clichy
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Compiegne, Compiègne
  - Centre Hospitalier Sud Francilien - Site Corbeil, Corbeil
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Du Bocage, Dijon
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - Institut Prive de Cancerologie, Grenoble
  - Centre Hospitalier, Juvisy-sur-Orge
  - Hopital Andre Mignot, Le Chesnay
  - C.H.G. Du Havre - Hopital J. Monod, Le Havre
  - Centre Hospitalier Universitaire de Bicetre, Le Kremlin-Bicêtre
  - Clinique Victor Hugo, Le Mans
  - Centre Hospitalier Lens, Lens
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Hospitalier General, Lons-le-Saunier
  - Clinique Saint Jean, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - Hopital Notre-Dame de Bon Secours, Metz
  - Intercommunal Hospital, Montfermeil
  - Clinique Gui de Chauliac, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Hopital Pasteur, Nice
  - Centre Antoine Lacassagne, Nice
  - C.H.U. de Nimes - Groupe Hospitals-Universitaire Caremeau, Nîmes
  - Hopital Saint Antoine, Paris
  - Hopital de la Croix Rouge Francaise des Peupliers, Paris
  - Hotel Dieu de Paris, Paris
  - Institut Curie - Section Medicale, Paris
  - Hopital Lariboisiere, Paris
  - Hopital Saint-Louis, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Cochin, Paris
  - Hopital Necker, Paris
  - C.H.G. De Pau, Pau
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Intercommunal de Poissy, Poissy
  - Hopital Rene Dubos, Pontoise
  - Polyclinique De Courlancy, Reims
  - CHG Roanne, Roanne
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - C.H.U. Saint Etienne Hospital Nord, Saint-Etienne
  - Hopital de Saint Germain-en-Laye, Saint-Germain-en-Laye
  - Centre Medico-Chirurgical Foch, Suresnes
  - Centre Hospitalier Regional de Purpan, Toulouse
  - Centre Hospitalier Valence, Valence
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - CHU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedale Sta. Maria Delle Croci, Ravenna
  - Ospedale S. Giovanni A.S. Dipartimente di Oncologia di Turin, Turin
- Netherlands (24):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Medisch Centrum Alkmaar, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - Comprehensive Cancer Center Amsterdam, Amsterdam
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Streekziekenhuizen Gooi-Noord, Blaricum
  - Amphia Ziekenhuis - locatie Molengracht, Breda
  - Atrium Medisch Centrum - Brunssum, Brunssum
  - Reinier de Graaf Group, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Academisch Ziekenhuis Groningen, Groningen
  - Atrium Medical Centre, Heerlen
  - Radiotherapeutisch Instituut, Leeuwarden
  - Diaconessenhuis Leiden, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Sint Antonius Ziekenhuis, Nieuwegein
  - University Medical Center Nijmegen, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - Maasland Hospital, Sittard
  - Leyenburg Ziekenhuis, The Hague
  - Academisch Ziekenhuis Utrecht, Utrecht
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Instituto Portugues de Oncologia Centro do Porto, SA, Porto, Portugal
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Institute of Oncology, Ljubljana, Ljubljana, Slovenia
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Switzerland (2):
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne

REFERENCES:
- [Background] van der Kaaij MA, Heutte N, van Echten-Arends J, Raemaekers JM, Carde P, Noordijk EM, Ferme C, Thomas J, Eghbali H, Brice P, Bonmati C, Henry-Amar M, Kluin-Nelemans HC. Sperm quality before treatment in patients with early stage Hodgkin's lymphoma enrolled in EORTC-GELA Lymphoma Group trials. Haematologica. 2009 Dec;94(12):1691-7. doi: 10.3324/haematol.2009.009696. Epub 2009 Oct 22. PMID 19850901
- [Background] van der Kaaij MA, Heutte N, Le Stang N, Raemaekers JM, Simons AH, Carde P, Noordijk EM, Ferme C, Thomas J, Eghbali H, Kluin-Nelemans HC, Henry-Amar M; European Organisation for Research and Treatment of Cancer: EORTC Lymphoma Group; Groupe d'Etude des Lymphomes de l'Adulte. Gonadal function in males after chemotherapy for early-stage Hodgkin's lymphoma treated in four subsequent trials by the European Organisation for Research and Treatment of Cancer: EORTC Lymphoma Group and the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2007 Jul 1;25(19):2825-32. doi: 10.1200/JCO.2006.10.2020. Epub 2007 May 21. PMID 17515571
- [Result] Eghbali H, Brice P, Creemers GY, et al.: Comparison of three radiation dose levels after EBVP regimen in favorable supradiaphragmatic clinical stages (CS) I-II Hodgkin's lymphoma (HL): preliminary results of the EORTC-GELA H9-F trial. [Abstract] Blood 106 (11): A-814, 2005.
- [Result] Ferme C, Diviné M, Vranovsky A, et al.: Four ABVD and involved-field radiotherapy in unfavorable supradiaphragmatic clinical stages (CS) I-II Hodgkin's lymphoma (HL): preliminary results of the EORTC-GELA H9-U trial. [Abstract] Blood 106 (11): A-813, 2005.
- [Result] Girinsky T, Gargi T, Carrie C, et al.: Quality assurance program in the EORTC-GELA H9 randomized study results on 282 patients. [Abstract] Int J Radiat Oncol Biol Phys 63 (2 Suppl 1): A77, S47, 2005.
- [Result] Noordijk EM, Thomas J, Fermé C, et al.: First results of the EORTC-GELA H9 randomized trials: the H9-F trial (comparing 3 radiation dose levels) and H9-U trial (comparing 3 chemotherapy schemes) in patients with favorable or unfavorable early stage Hodgkin's lymphoma (HL) . [Abstract] J Clin Oncol 23 (Suppl 16): A-6505, 561s, 2005.
- [Result] Thomas J, Ferme C, Noordijk EM, et al.: Six cycles of EBVP followed by 36 Gy involved-field irradiation vs. no irradiation in favourable supradiaphragmatic clinical stages I-II Hodgkin's lymphoma: the EORTC-GELA strategy in 771 patients (H9-F trial-20982). [Abstract] Eur J Haematol 75 (Suppl 65): A-E11a, 40, 2004.
- [Result] Thomas J, Ferme C, Noordijk EM, et al.: Six cycles of ABVD + IF-RT vs. four cycles of ABVD + IF-RT vs. four cycles of BEACOPP + IF-RT in unfavourable supradiaphragmatic clinical stages I-II Hodgkin's lymphoma: the EORTC-GELA H9-U randomized clinical trial (20982) in 808 patients. [Abstract] Eur J Haematol 73 (Supp 65): A-E12, 40, 2004.
- [Derived] Thomas J, Ferme C, Noordijk EM, Morschhauser F, Girinsky T, Gaillard I, Lugtenburg PJ, Andre M, Lybeert MLM, Stamatoullas A, Beijert M, Helias P, Eghbali H, Gabarre J, van der Maazen RWM, Jaubert J, Bouabdallah K, Boulat O, Roesink JM, Christian B, Ong F, Bordessoule D, Tertian G, Gonzalez H, Vranovsky A, Quittet P, Tirelli U, de Jong D, Audouin J, Aleman BMP, Henry-Amar M. Comparison of 36 Gy, 20 Gy, or No Radiation Therapy After 6 Cycles of EBVP Chemotherapy and Complete Remission in Early-Stage Hodgkin Lymphoma Without Risk Factors: Results of the EORT-GELA H9-F Intergroup Randomized Trial. Int J Radiat Oncol Biol Phys. 2018 Apr 1;100(5):1133-1145. doi: 10.1016/j.ijrobp.2017.10.015. Epub 2017 Oct 27. PMID 29229324
- [Derived] Ferme C, Thomas J, Brice P, Casasnovas O, Vranovsky A, Bologna S, Lugtenburg PJ, Bouabdallah R, Carde P, Sebban C, Eghbali H, Salles G, van Imhoff GW, Thyss A, Noordijk EM, Reman O, Lybeert MLM, Janvier M, Spina M, Audhuy B, Raemaekers JMM, Delarue R, Anglaret B, de Weerdt O, Marjanovic Z, Tersteeg RJHA, de Jong D, Briere J, Henry-Amar M; European Organisation for Research and Treatment of Cancer Lymphoma Group, and; Groupe d'Etude des Lymphomes de l'Adulte. ABVD or BEACOPPbaseline along with involved-field radiotherapy in early-stage Hodgkin Lymphoma with risk factors: Results of the European Organisation for Research and Treatment of Cancer (EORTC)-Groupe d'Etude des Lymphomes de l'Adulte (GELA) H9-U intergroup randomised trial. Eur J Cancer. 2017 Aug;81:45-55. doi: 10.1016/j.ejca.2017.05.005. Epub 2017 Jun 8. PMID 28601705